CLINICAL TRIAL: NCT02244190
Title: Bioequivalence of Two Different Oral Solutions of 500 mg of Tipranavir (New Formulation vs. Current Formulation) Administered in Combination With 200 mg of Ritonavir (Oral Solution) to Healthy Volunteers (an Open-label, Randomised, Single Dose, Two-way Crossover Study)
Brief Title: Bioequivalence of Two Different Oral Solutions Tipranavir Administered in Combination With Ritonavir to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1182.124
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir

ARMS (2):
- new Tipranavir + Ritonavir (Experimental)
  Interventions: Drug: Tipranavir; Drug: Ritonavir
- current Tipranavir + Ritonavir (Active Comparator)
  Interventions: Drug: Tipranavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Tipranavir — New oral solution (back up) formulation
  Arms: new Tipranavir + Ritonavir
Drug: Tipranavir
  Other Names: Current oral solution formulation
  Arms: current Tipranavir + Ritonavir
Drug: Ritonavir
  Other Names: Norvir®

SUMMARY:
To establish the bioequivalence of the new tipranavir oral solution formulation with the current tipranavir oral solution formulation following single-dose administration. In each case, 500 mg tipranavir was coadministered with 200 mg ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2 (Body Mass Index) and body weight > 55 kg
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to tipranavir or ritonavir or their excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration of the trial drug or during the trial
* Cytochrome P 450 (CYP3A4)-inhibiting drugs (e.g. itraconazole, ketoconazole, protease inhibitors, erythromycin, clarithromycin, telithromycin, nefazodone, cyclosporin, verapamil, amiodarone, diltiazem), CYP3A4 inducing drugs (e.g. St. John´s wort [Hypericum perforatum], rifampin, dexamethasone) or CYP3A4 substrates (e.g. triazolam, sertraline); further drugs which might reasonably influence the results of the trial (e.g. drugs which contain polyethylene glycol) or drugs that prolong the QT/corrected QT interval interval (based on the knowledge at the time of protocol preparation) within 14 days prior to first administration of the trial drug or during the trial
* Participation in another trial with an investigational drug within two months prior to administration of the trial drug or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking within 24 hours before or after administration of the trial drug
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration of the trial drug or during the trial)
* Excessive physical activities (within one week prior to administration of the trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de Pointes (TdP), e.g., heart failure, hypokalaemia, family history of Long QT Syndrome
* Known hypersensitivity to antiretroviral drugs (marketed or experimental use as part of clinical research studies)
* Personal or family history of coagulation or bleeding disorders or bleeding tendencies
* Intake of vitamin E within 14 days prior to the first drug administration of this trial or during the trial
* Transaminase values (ALT /AST) greater than the upper limit of the normal laboratory reference range during screening

For female subjects:

* Pregnancy or positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
* No adequate contraception during the study and until 1 month of study completion, i.e. not any of the following: implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females who do not have a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide).
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of drug in plasma over the time interval from 0 extrapolated to infinity) for tipranavir | up to 72 hours after drug administration
Cmax (maximum measured concentration of drug in plasma) for tipranavir | up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ for ritonavir | up to 72 hours after drug administration
Cmax for ritonavir | up to 72 hours after drug administration
AUC0-tz (area under the concentration-time curve of drug in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of drug in plasma) | up to 72 hours after drug administration
λz (terminal rate constant of drug in plasma) | up to 72 hours after drug administration
t1/2 (terminal half-life of drug in plasma) | up to 72 hours after drug administration
MRTpo (mean residence time of drug in the body after oral administration) | up to 72 hours after drug administration
CLpo/F (apparent clearance of drug after oral administration) | up to 72 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours after drug administration
Number of patients with adverse events | up to 43 days
Number of patients with clinically significant findings in vital signs | up to 43 days
Number of patients with clinically significant findings in 12-lead electrocardiogram | up to 43 days
Number of patients with clinically significant findings in laboratory tests | up to 43 days
Assessment of tolerability by investigator on a 4-point scale | Day 4 of each treatment period